CLINICAL TRIAL: NCT01992744
Title: Peripheral Serum BDNF Levels and Poor Birth Outcomes
Brief Title: BDNF Pregnancy Study
Acronym: BDNF
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 815839
Record Dates: First submitted 2013-10-30; First posted 2013-11-25 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2013-10

CONDITIONS: Pregnancy
Keywords: pregnancy; brain-derived neurotrophic factor; birth outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — - Brain-Derived Neurotrophic Factor
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy Pregnant Women: Participants 8 to 12 weeks gestational age as determined by their physician.

SUMMARY:
The purpose of this study is to evaluate the correlation between varying levels of neuropeptides and birth outcomes. Neuropeptides are substances (proteins) produced in the body in very small amounts but without which the nervous system cannot function properly, and which might have a role in the health of a newborn. As part of this study, we are collecting blood samples from pregnant women.

Neuropeptides and hormones can be measured in blood. This study will involve three blood draws from the participants arm. Demographic information will also be requested, and participants will be asked to complete questionnaires about their mood and personal experiences at each visit.

Our hypothesis is that participants with lower levels of brain-derived neurotrophic factor (BDNF) will be at increased risk for poor birth outcomes.

DETAILED DESCRIPTION:
This prospective, non-randomized trial will evaluate peripheral serum blood levels of BDNF in participants recruited from previously identified University of Pennsylvania obstetrics and gynecological (OB/GYN) clinics. A total of 100 pregnant subjects will be recruited consecutively and evaluated in the first and third trimester of their pregnancy as well as within a month after delivery.

The entire project will take one year.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at least 18 years old and being treated at an outpatient OB/GYN clinic;
* At least 8 weeks pregnant;
* Capable of giving informed consent.

Exclusion Criteria:

* Participants younger than 18 years of age;
* History of preterm birth;
* Psychiatric medications during current pregnancy;
* Participants with a history of hematologic disorders;
* Participants who refuse informed consent.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women from the greater Philadelphia and surrounding areas who are ages 18 to 39 and between 8 to 12 weeks pregnant will be considered for enrollment into this study. All subjects must be physically healthy without a serious, major medical illness as well as be carrying a healthy fetus. Subject will be enrolled through OB/GYN waiting room recruiting, fliers, advertisements and social media outlets.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2012-05; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Neuropeptide & Blood Levels | First Trimester (8 weeks to 12 weeks gestational age), Third Trimester (28 weeks to 32 weeks gestational age) & Postpartum (30 days postpartum)
  * BDNF
  * Complete blood count (CBC)

SECONDARY OUTCOMES:
Clinician and Patient Ratings | First Trimester (8 weeks to 12 weeks gestational age), Third Trimester (28 weeks to 32 weeks gestational age) & Postpartum (30 days postpartum)
  * Edinburgh Postnatal Depression Score (EPDS)
  * Perceived Stress Scale Score (PSS)
  * Adverse Childhood Events Questionnaire Score (ACEs)
  * Beck Depression Inventory (BDI)
  * Brief Anxiety Inventory (BAI)
  * Brief Symptom Inventory (BSI)

OTHER OUTCOMES:
Birth Outcomes | Postpartum (30 days postpartum)
  * Birth weight (low birth weight < 2.5 kg; very low birth weight < 1.5 kg)
  * APGAR score (at one minute, at five minutes)
  * Preterm birth (before 37 weeks gestation; very early preterm birth, before 35 weeks gestation); gestational age at delivery
  * Infant mortality/ Neonatal Intensive Care Unit (NICU) Admission
  * Major congenital malformations (especially neurologic)
  * Head circumference (cm)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah R Kim, M.D., Principal Investigator — Assistant Professor University of Pennsylvania
Locations (4):
- United States (4):
  - 3701 Market Street, Philadelphia, Pennsylvania
  - Helen O. Dickens Center for Women's Health, Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Penn Center for Women's Behavioral Wellness, Philadelphia, Pennsylvania
  - Penn Medicine Washington Square (PMWS), Philadelphia, Pennsylvania

REFERENCES:
- [Background] Kim DR, Gonzalez JM, Sammel MD, Parry S, Epperson CN. Brain Derived Neurotrophic Factor is Altered in Human Pregnancy. Clinical Neuropsychiatry 2012 Dec; 9(6):207-11.
- See also: Program Website — http://www.med.upenn.edu/womenswellness/